CLINICAL TRIAL: NCT04856215
Title: 90Yttrium-labelled Anti-CD66 Monoclonal Antibody as Part of a Reduced Toxicity Conditioning Regimen Prior to Allogeneic Haematopoietic Stem Cell Transplantation: an Open Label, Phase II Study in Children and Adolescents With High Risk Leukaemia
Brief Title: 90Y-labelled Anti-CD66 ab in Childhood High Risk Leukaemia
Acronym: RITII
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17WA58
Record Dates: First submitted 2021-04-13; First posted 2021-04-23 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 90-Yttrium-labelled anti-CD66 monoclonal antibody (Experimental): The medicinal product consists of the murine IgG1 anti-CD66 monoclonal antibody radio-labelled with 111In for imaging and dosimetry and with 90Y for therapy.
  Dosage indications The [111In]-labeled anti-CD66 monoclonal antibody (MAb) will be given at an infused activity of 100MBq/sqm between 1-4 weeks before the therapeutic dose of radiolabelled antibody.
  [90Y]-yttrium-labeled anti-CD66 MAb will be given as a single infusion on day - 14 prior to transplant. [90Y]-yttrium labelled anti-CD66 MAb will be given to target an absorbed dose to the bone marrow of 45 Gy +/- 10%. The maximum dose to be delivered to the liver and the kidneys is 15 Gy and 10 Gy, respectively.
  Interventions: Drug: 90-Yttrium-labelled anti-CD66 monoclonal antibody

INTERVENTIONS:
Drug: 90-Yttrium-labelled anti-CD66 monoclonal antibody — The Investigational Medicinal Product (IMP) consist of 1) 111Indium- and 2) 90Yttrium-labelled anti-CD66 (BW250/183) monoclonal antibody.
  The anti-CD66 is a murine IgG1 monoclonal antibody originally developed as an in vivo leucocyte and bone marrow imaging agent (Boßlet 1985, Thomsen 1991). BW 250/183 anti-CD66 is a murine IgG1 kappa monoclonal antibody, originally produced as an anti-CEA antibody.
  The batch of antibodies required for treatment will be radiolabelled by Royal Free Hospital radiology team with Indium 111 and Y90 for patient.

SUMMARY:
Children affected by high risk or relapsed/refractory leukaemia have a poor prognosis, with an increased risk of relapse. These patients generally need treatment intensification and a bone marrow transplantation (BMT).

Nevertheless, with conventional treatent the risk of relapse after transplant remains high.

Radioimmunotherapy provides a way to deliver high dose irradiation to the bone marrow (where leukaemia resides), while sparing normal organs and tissues from its toxicity.This can be achieved by linking a radioactive molecule (Yttrium90) to an antibody that, once infused in the blood, targets marrow/leukemic cells.

DETAILED DESCRIPTION:
In our Phase 1 trial which concluded in 2019, 9 children affected by refractory or relapsed leukaemia were enrolled at Great Ormond Street Hospital or UCLH. Participants received infusion of a tumour cell targeting antibody to deliver irradiation to the bone marrow and sites containing leukemic blasts prior to BMT. The aim of the Phase 1 study was to identify the dose limiting toxicity and maximum tolerated dose of targeted radiotherapy, and it was found that this treatment was well tolerated with minimal infusion-related side effects.

The current study will enrol a larger cohort of children (aged 0.5 - 18 years) who will receive 90Yttrium administered at an infused activity to target the optimal absorbed dose to the bone marrow. Patients will be treated at GOSH and UCLH and followed up for 12 months post-BMT to evaluate safety and efficacy of targeted radiotherapy with a reduced toxicity conditioning regimen prior to BMT.

PURPOSE AND DESIGN OF THE STUDY Children with high risk or relapsed leukaemia have a poor prognosis with an increased risk of relapse after standard bone marrow transplant. There is an urgent need to offer a different therapeutic strategy for children with such poor risk diseases.

There is evidence that targeted radioimmunotherapy prior to a stem cell transplantation is a feasible and effective treatment that delivers high dose radiation to the bone marrow and spleen (where leukaemia resides),while sparing other tissues and organs from its toxicity. Since leukaemic cells are generally radiosensitive, this approach might increase leukaemia-free survival, while reducing transplant-related morbidity and mortality.

Our previous phase 1 radio-immunotherapy study demonstrated that radio-immunotherapy is non-toxic, but can elicit myelosuppression, with potential for better disease eradication.

This protocol offers a novel and non-toxic therapeutic strategy to children with poor risk leukaemia and aims at reducing the risk of disease relapse after transplant.

RECRUITMENT and CONSENT Children with poor risk leukaemia who fulfill the inclusion and exclusion criteria of this study might be recruited in this trial. Patients and/or their parents will receive appropriate information from one of the investigators regarding the rationale of this study, the possible risks and benefits and the alternatives to taking part. Patients and/or their parents will be given an age appropriate information sheet and consent form and they will be given the time to think about this.

INCLUSION/EXCLUSION CRITERIA Children enrolled in this study must be affected by high risk or relapsed/refractory leukaemia, with a high risk of disease relapse after conventional transplant. Children eligible for this treatment must also be clinically fit for an allogeneic haematopoietic stem cell transplantation, according to clinical and laboratory parameters, which have been specified in details in the protocol.

RISKS, BURDENS AND BENEFITS Patients eligible for this trial are affected by high risk or relapsed/refractory leukaemia and have an indication to an allogeneic stem cell transplantation. Stem cell transplantation carries a significant risk of morbidity/mortality, due to: a)the toxicity of the preparative regimen, b) the posttransplant immunodeficiency with high risk of opportunistic infections, and c) the possible occurrence of graft versus host disease. The use of radioimmunotherapy in the context of a reduced toxicity conditioning regimen prior to the transplantation has proved to be feasible and safe in adult and paediatric studies, without a significant increase of the treatment related toxicity when compared to standard conditioning regimen.

Moreover, higher doses of radiation delivered to patients with leukaemia generate a better leukaemia response and this approach in children with poor risk leukaemia is promising.

Children undergoing this treatment will be carefully followed up and haematological (prolonged cytopaenia, stromal damage) and nonhaematological (mucositis, liver and kidney damage)toxicity will be monitored and recorded.

ELIGIBILITY:
Inclusion Criteria:

1. An underlying hematological malignancy including:

   a) relapse of AML after allogeneic hematopoietic stem cell transplantation; b) relapse of ALL after allogeneic hematopoietic stem cell transplantation; c) relapse of JMML after allogeneic hematopoietic stem cell transplantation; e) refractory ALL; f) refractory AML; g) high risk infant ALL;
2. be ≥ 0.5 year old and ≤ 18 years old;
3. must not be eligible for therapy of higher curative potential. Where an alternative therapy has been shown to prolong survival in an analogous population, this should be offered to the patient prior to discussing this study;
4. have a Karnofsky Performance Status ≥ 50 or Lansky Performance Status ≥ 30;
5. provide signed, written informed consent from parent or guardian;
6. be able to comply with study procedures and follow-up examinations;
7. have adequate cardiac function (irrespective of concomitant cardio-vascular treatment) at PI/CI discretion;
8. have adequate organ function (as indicated by Table 5) within 30 days prior to 111In infusion;
9. patients who have received any other chemotherapy within the previous 2 weeks and must have recovered from acute toxicity of all previous therapy prior to enrolment;
10. be negative for human-anti-murine antibodies (HAMA).

Exclusion Criteria:

1. patients who are positive for human anti-murine antibodies (HAMA);
2. patients with compromised organ function within 30 days prior to 111In infusion;
3. patients with isolated CNS disease relapse*;
4. patients with an active, uncontrolled systemic infection considered opportunistic, life threatening, or clinically significant at the time of treatment;
5. Pregnant or breast-feeding females are excluded due to potential risks of foetal adverse events of an investigational agent. Pregnancy tests must be obtained prior to enrolment on this study for girls of reproductive potential. The need to commence pregnancy testing will be at the discretion of the treating physician to facilitate taking in to account factors such as precocious puberty, endocrine status and medications which can affect pubertal status. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method. Sexual Abstinence is an acceptable method of birth control**.
6. patients with any other severe concurrent disease, which, in the judgment of the Investigator, would make the patient inappropriate for entry into this study;
7. patients with extensive chronic graft versus host disease (GVHD);
8. patients with unstable cardio-vascular disease. -

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Disease response after [90Y]-labelled anti-CD66 monoclonal antibody | through study completion, upto 2 years post study
  recovery of normal hematopoiesis in the bone marrow, with blasts < 5% of lymphoid/myeloid cells and lack of evidence for residual leukemia using any informative cytogenetic/molecular marker. The number and proportion of patients who have a response will be provided in each cohort.

SECONDARY OUTCOMES:
Assessment of timing of myeloid and platelet engraftment after allogeneic hematopoietic stem cell transplantation. | through study completion, upto 2 years post study
  Assessment of timing of myeloid and platelet engraftment after allogeneic hematopoietic stem cell transplantation.
Assessment of chimerism on bone marrow and peripheral blood to confirm engraftment of donor origin. | through study completion, upto 2 years post study
  Assessment of chimerism on bone marrow and peripheral blood to confirm engraftment of donor origin.
Safety Outcome | through study completion, upto 2 years post study
  Toxicity will be classified using the National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Chiesa, Principal Investigator — Great Ormond Street Hospital
Locations (2):
- United Kingdom (2):
  - Great Ormond Street Hospital NHS Foundation Trust, London
  - University College London Hospital NHS Trust, London

IPD SHARING:
Plan to Share IPD: No